CLINICAL TRIAL: NCT02263755
Title: Establishment of Retrospective and Prospective Multicenter Cohort for Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0582
Record Dates: First submitted 2014-09-03; First posted 2014-10-13 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Hepatitis B
Keywords: CHB, cohort, fibroscan
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- chronic hepatitis B subjects: Subjects who have been diagnosed with chronic hepatitis B.

SUMMARY:
According to the World Health Organization about 1,400,000 deaths reported annually, are related to chronic liver disease. Chronic liver disease is very prevalent in South Korea, placing a large economic burden nationwide. Subsequently, an effective and systematized approach to managing chronic hepatitis is imperative in Korea.

The natural history of chronic liver disease differs greatly according to race and ethnicity. However, there is scarcity of epidemic data on chronic hepatitis based on Korean patients. Therefore, the investigators plan to establish a retrospective and prospective multicenter cohort for chronic hepatitis B based on Korean patients that may be utilized for various future clinical studies on chronic hepatitis B in Korea, and thereby serve as a basis for the establishment and distribution of clinical guidelines for Korean patients with chronic hepatitis B, as part of a nationwide project supported by the Centers for Disease Control (CDC), Korea.

The investigators plan to collect 500 cases as have been advised by the CDC during the study period (September, 2014-March, 2015) from 4 tertiary hospitals located in Korea. In the past 5 years, there have been about 800 subjects with chronic hepatitis B who have undergone liver fibroscan and liver biopsy from these 4 institutions. The investigators plan to register available cases retrospectively from those who are available to agree to give written informed consent to participate in this study, and to register the remaining numbers of cases prospectively, according to the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Subject aged 20 years or older
2. Subject who has been diagnosed with chronic hepatitis B (HBs Ag (+) for minimum of 6 months_
3. Subject who is currently under clinical follow up at the registered institution
4. Subject who has undergone or who can undergo liver fibroscan at the time of registration
5. Subject who has given informed consent to the enrollment

Exclusion Criteria:

1. Subject with decompensated liver cirrhosis or hepatocellular carcinoma at the time of initial liver fibroscan
2. Subject who had previously undergone antiviral therapy for chronic hepatitis B
3. Subject who are concomittantly infected with HCV, HDV or HIV
4. Subject with chronic alcoholism defined as equal to or greater than 40g of alcohol for duration of 5 years or longer
5. Subject who has been diagnosed with right sided heart failure
6. Subjects whose liver fibroscan result is not valid
7. Subject who is considered ineligible to the enrollment to clinical study by the researcher
8. Subjects who is pregnant at the time of registration
9. Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatient clinic in tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 476 (Actual)
Dates: Start 2014-09-02 (Actual); Primary Completion 2015-06-25 (Actual); Study Completion 2015-06-25 (Actual)

PRIMARY OUTCOMES:
retrospective and prospective multicenter cohort for chronic hepatitis B based on Korean patients | time of registration of patient to cohort completment
  This study aims for the establishment of chronic hepatitis B cohort and has no other primary end point other than the registration of the patient. (For Time-to-Event outcome measures, the development of events including HCC, ascitic decompensation, variceal bleeding, hepatic encephalopathy, transplantation, and death will be followed up to 10 years after enrollment. Time to the development of each kind of event will be calculated from the date of enrollment and the respective date of event development.)

CONTACTS AND LOCATIONS:
Overall Officials: Kwang Hyub Han, MD,PhD, Principal Investigator — Yonsei University

REFERENCES:
- [Background] Jung KS, Kim SU, Ahn SH, Park YN, Kim DY, Park JY, Chon CY, Choi EH, Han KH. Risk assessment of hepatitis B virus-related hepatocellular carcinoma development using liver stiffness measurement (FibroScan). Hepatology. 2011 Mar;53(3):885-94. doi: 10.1002/hep.24121. Epub 2011 Feb 11. PMID 21319193
- [Background] Kim SU, Ahn SH, Park JY, Kang W, Kim DY, Park YN, Chon CY, Han KH. Liver stiffness measurement in combination with noninvasive markers for the improved diagnosis of B-viral liver cirrhosis. J Clin Gastroenterol. 2009 Mar;43(3):267-71. doi: 10.1097/MCG.0b013e31816f212e. PMID 18987556
- [Background] Kim SU, Seo YS, Cheong JY, Kim MY, Kim JK, Um SH, Cho SW, Paik SK, Lee KS, Han KH, Ahn SH. Factors that affect the diagnostic accuracy of liver fibrosis measurement by Fibroscan in patients with chronic hepatitis B. Aliment Pharmacol Ther. 2010 Aug;32(3):498-505. doi: 10.1111/j.1365-2036.2010.04353.x. Epub 2010 May 11. PMID 20491742